CLINICAL TRIAL: NCT06832449
Title: Retrospective Clinical Trial Investigating the Treatment of Chronic Pain With the Freedom Peripheral Nerve Stimulation System
Brief Title: Retrospective PNS Study
Status: Active, not recruiting | Type: Observational
Sponsor: Curonix LLC (Industry)
Collaborators: Colorado pain Care, LLC (Unknown)
Responsible Party: Sponsor
Other Study IDs: P017
Record Dates: First submitted 2025-02-11; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Chronic Pain
Keywords: Retrospective, chronic pain, PNS
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: PNS — Retrospective study investigating PNS

SUMMARY:
Retrospective PNS Study

ELIGIBILITY:
Inclusion Criteria:

A. Subjects are at least 18 years of age, B. Subjects have been diagnosed with refractory chronic pain, C. Subject has been implanted with a permanent Freedom Peripheral Nerve Stimulation System.

Exclusion Criteria:

A. Any additional active implanted devices for the treatment of chronic pain in addition to the Freedom Peripheral Nerve Stimulation System.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 200
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
VRS | 36 months
  A text description of the subject's pain location(s) and severity will be recorded to correlate with subject feedback. The VRS will be used to measure severity.

SECONDARY OUTCOMES:
Health economic data | 12 months
  The value of claims data at the site will be measured from 1 year before and up to the date of implant and compared to the claims value up to 1 year after implant. The number of appointments will be collected together with the CPT codes used for pain interventions.

CONTACTS AND LOCATIONS:
Locations (1):
- Colorado Pain Care, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided